CLINICAL TRIAL: NCT04708860
Title: Pilot Study of the Impact of a Combined Intermittent Fasting and Exercise Intervention on Metabolic Markers in Patients With Advanced, Hormone Receptor Positive Breast Cancer
Brief Title: Feasibility of Fasting & Exercise in Pts With HR+ MBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer A. Ligibel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-503
Record Dates: First submitted 2021-01-04; First posted 2021-01-14 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
Keywords: Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolonged Nightly Fasting Plus Exercise (Experimental): Participants will be grouped into two cohorts determined by whether they receive palbociclib or alpelisib as part of their breast cancer treatment and then receive a 12 week prolonged nightly fasting plus exercise program consisting of:
  * Prolonged overnight fasting: Not consume any calorie-containing food/drinks after 8pm, waiting a minimum of 13 hours after their last meal of the day before eating the next day, target goal of fasting at least 6 days a week, daily record of first and last meals
  * Exercise Program: Coach provided at-home, personalized exercise regimen with target goal of 120 minutes of moderate-intensity aerobic activity each week as well as two 30-45-minute virtual strength training classes per week, receive fitbit for exercise and heart rate monitoring, weekly telephone-based support sessions with coach.
  Interventions: Behavioral: Prolonged Nightly Fasting; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Prolonged Nightly Fasting — Restriction of consumption of calorie-containing food/drinks after 8pm
Behavioral: Exercise — Personalized moderate-intensity, aerobic exercise and strength training

SUMMARY:
This research is evaluating the impact of a 12-week prolonged nightly fasting (POF) and exercise intervention on metabolic markers and patient reported outcomes in women with metastatic breast cancer (MBC) initiating endocrine therapy in combination with palbociclib or alpelisib.

DETAILED DESCRIPTION:
This is single-arm feasibility pilot study exploring whether a combined prolonged nightly fasting (POF) and exercise program could impact hyperglycemia and other adverse metabolic consequences of PI3 kinase inhibitors in women with metastatic breast cancer (MBC).

Women who exercise regularly and who have lower levels of blood sugar and metabolic hormones like insulin have a lower risk of developing breast cancer. Some evidence also suggests that exercise and metabolism are related to cancer recurrence in women who are diagnosed with breast cancers that can be removed with surgery, but less is known about how exercise and metabolic factors are related to cancer progression in women whose cancer has advanced beyond the breast and underarm lymph nodes. This study is designed to look at the effects of exercise combined with prolonged nightly fasting (having a longer time between dinner and breakfast the next day), on blood sugar and hormones that control metabolism. This study looks to provide important information about whether making these kinds of changes is possible for women living with advanced breast cancer and will explore how making these changes effects blood sugar and hormone levels in women taking different kinds of treatments for advanced breast cancer.

The research study procedures include screening for eligibility, a baseline visit to collect information about diet and exercise habits, a baseline blood draw, participation in a 12-week diet and exercise program, and a follow up visit and blood collection at the end of the diet and exercise program.

Participants will be in this research study for up to 14-weeks, including the baseline and end of study visits to collect study measures.

It is expected that about 30 people will take part in this research study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ER and/or PR+ metastatic or locally unresectable breast cancer
* Postmenopausal (including concurrent use of ovarian suppression)
* Initiating endocrine therapy in combination with:

  * Cohort 1: alpelisib
  * Cohort 2: palbociclib
* Self-reported ability to walk two blocks
* > 18 years of age
* Approval from treating oncologist, confirmed via email or in writing
* Ability to read and understand English

Exclusion Criteria:

* Diagnosis of diabetes requiring medication
* Engaging in >90 minutes of moderate or vigorous physical activity per week

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of enrollment | 12 months
  The primary objective is to evaluate the feasibility of the intervention. Feasibility will be defined by the rate of enrollment and the intervention will be considered feasible if at least 80% of planned participants are enrolled within 12 months of study activation.
Rate of adherence to prolonged overnight fasting (POF) intervention goals | 12 weeks
  Feasibility will additionally be defined by participants achieving POF intervention goals on 70% of days by week 12.
Rate of adherence to exercise intervention goals | 12 weeks
  Feasibility will also be defined by at least 70% of participants achieving 120 minutes of aerobic exercise plus 2 strength training classes per week by week 12.

SECONDARY OUTCOMES:
Changes in metabolic biomarkers between baseline and week 12 | 12 weeks
  We will evaluate changes in fasting glucose, insulin, insulin resistance, hemoglobin A1c and other metabolic biomarkers in study participants between the baseline and end-of-intervention blood draws.
Change in quality of life and patient-reported outcome measures between baseline and week 12 | 12 weeks
  Quality of life will be evaluated for participants at baseline and at the end of the intervention using the EORTC QLQ C-30, sleep quality will be assessed via the Pittsburgh Sleep Quality Index (PSQI). Additional patient reported outcomes include the PRO-CTCAE, the 7-Day Physical Activity Recall and the 24-Hour Dietary Recall. We will assess changes in these measures between baseline and week 12 for study participants.
Differences in changes in metabolic biomarkers by treatment group (palbociclib vs palbocilib) | 12 weeks
  We will explore potential differences in changes in metabolic markers over the course of the 12-week POF and exercise intervention by treatment group (alpelisib vs palbociclib).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ligibel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu